CLINICAL TRIAL: NCT06033248
Title: Validation and Determination of Feasibility for Clinical Use of an Animal Biosensor Platform to Detect Non-Small Cell Lung Cancer-Specific Volatile Organic Compounds in Urine Samples
Brief Title: Using Urine Samples to Identify Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: EARLY Labs (Unknown)
Responsible Party: Sponsor
Other Study IDs: 23-111
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Urine samples; stages I, II, and IIIA; 23-111
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients diagnosed with NSCLC: In phase I, the researchers will assess the ability of a rat-based ABP to detect the presence or absence of NSCLC-specific VOCs in urine samples from subjects with and without NSCLC. In phase II, the researchers will assess the ability of the ABP to detect the presence of NSCLC-specific VOCs in urine samples from subjects with suspected but undiagnosed NSCLC (clinical stage I to IIIA). Urine samples will be collected from 50 patients diagnosed with NSCLC and from 50 subjects without NSCLC for phase I and from 110 patients with suspected but undiagnosed NSCLC for phase II (total number of subjects = 210).
  Interventions: Diagnostic Test: urine sample

INTERVENTIONS:
Diagnostic Test: urine sample — urine sample will be collected

SUMMARY:
The researchers are doing this study to test the ability of an animal biosensor platform (ABP) to detect NSCLC. Participants in this study will either be diagnosed with NSCLC, suspected to have NSCLC, or have not been diagnosed or suspected to have NSCLC.

The ABP test uses laboratory animals that are trained to detect (by smell) different chemicals in urine. Studies show that people with lung cancer have unique chemicals in their urine that are not present in people without lung cancer, and researchers think these chemicals can be used to identify people with lung cancer without the need for invasive procedures (like biopsy).

ELIGIBILITY:
Inclusion Criteria:

* Phase I (with NSCLC): Aged 18 to 90 years with histologically proven, previously untreated stage I, II, or IIIA NSCLC

  °Note: Single, monolateral nodule of at least 50% solid composition visible on a Chest CT scan that is suspicious for a primary neoplasm as confirmed by an official MSK radiologist read
* Phase I (without NSCLC): Aged 18 to 90 years with patient confirmed absence of NSCLC
* Phase II: Aged 18 to 90 years with suspected but undiagnosed stage I, II, or IIIA NSCLC by CT and/or PET scan criteria

Exclusion Criteria:

* Aged <18 years
* Lack of available results from low-dose CT
* Receipt of radiation, chemotherapy, biological therapy, resection, or any other treatment for any cancer in the previous year
* Pregnant (for women)
* Taking drugs that affect the immune system
* Chronic disease related to the immune system
* Missing clinical data (i.e., current clinical staging)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thoracic Surgery clinics
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
detect the presence or absence of NSCLC-specific VOCs | 2 years
  in urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Rocco, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm